CLINICAL TRIAL: NCT07403552
Title: A Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of NSHO-101 in Healthy Participants
Brief Title: Evaluate the Pharmacokinetics, Safety, and Tolerability of NSHO-101 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ensho Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NSHO-101-HV202
Record Dates: First submitted 2026-01-26; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: To evaluate pharmacokinetics and safety of NSHO-101
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NSHO-101 Dose A (Experimental): Oral dose A of NSHO-101 QD for 14 days
  Interventions: Drug: NSHO-101
- NSHO-101 Dose B (Experimental): Oral dose B of NSHO-101 QD for 14 days
  Interventions: Drug: NSHO-101

INTERVENTIONS:
Drug: NSHO-101 — Dose form - tablet Route of administration - oral Regimen / Treatment period - QD for 14 days

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety, and tolerability of NSHO-101 in Healthy Participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants (males and females) at least 18 years of age
* Ability to provide written informed consent
* In good heath as determined by medical evaluation,
* Willing and able to comply with trial restrictions, procedures, and requirements

Exclusion Criteria:

* Known sensitivity to any components of the IMP
* History of relevant drug hypersensitivity
* Presents or has a history of clinically significant diseases
* History of difficulty swallowing tablets or capsules.
* Any physical examination findings or medical history that might place the participant at an unacceptable risk for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: Maximum Concentration (Cmax) | Day 1 to Day 18
Pharmacokinetics: Area Under the Concentration Curve (AUC) | Day 1 to Day 18
Pharmacokinetics: Trough Concentration (Ctrough) | Day 1 to Day 18
Pharmacokinetics: Half-life | Day 1 to Day 18
Pharmacokinetics: Time to Maximum Concentration (tmax) | Day 1 to Day 18

SECONDARY OUTCOMES:
Treatment Emergent Adverse Events | Day 1 to 14
  Incidence of TEAEs
Serious Treatment Emergent Adverse Events | Day 1 to Day 14
  Incidence of STEAEs

CONTACTS AND LOCATIONS:
Locations (1):
- Cenexel Anaheim CA, Anaheim, California, United States